CLINICAL TRIAL: NCT05444829
Title: Precision of Patient Specific Screw Holes Locating Surgical Guide and Pre-bent Plates Osteosynthesis Versus Classical Work-flow in Management of Class III Mandibular Fractures
Brief Title: Specific Screw Holes Locating Surgical Guide and Pre-bent Plates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abdallah Gaber Ali Mohamed (Other)
Responsible Party: Sponsor-Investigator, Abdallah Gaber Ali Mohamed, Researcher, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: class III mandibular fractures
Record Dates: First submitted 2022-06-22; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Mandibular Fractures
Keywords: class III
MeSH Terms: conditions — Mandibular Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- specific screw holes locating surgical guide and pre-bent plates (Experimental): Put the specific screw holes locating device in place and drill the screw holes, remove the screw holes locating device and mobilize the segments then apply the pre-bent plates and fix it with screw for passive reduction of the segments. Then suture the mentalis muscle then the mucosa.
  Interventions: Device: specific screw holes locating surgical guide and pre-bent plates
- classical reduction and fixation (Other): mobilize the broken segment first, Arch bar was made to achieve proper occlusion put the compression plate on the inferior border and remove it for further bending using plate pliers for further accommodation of the plate on the inferior border the fix it in place using compression and tension plate.
  Interventions: Device: classical reduction and internal fixation.

INTERVENTIONS:
Device: specific screw holes locating surgical guide and pre-bent plates — Put the specific screw holes locating device in place and drill the screw holes, remove the screw holes locating device and mobilize the segments then apply the pre-bent plates and fix it with screw for passive reduction of the segments. Then suture the mentalis muscle then the mucosa.
  Arms: specific screw holes locating surgical guide and pre-bent plates
Device: classical reduction and internal fixation. — mobilize the broken segment first, Arch bar was made to achieve proper occlusion put the compression plate on the inferior border and remove it for further bending using plate pliers for further accommodation of the plate on the inferior border the fix it in place using compression and tension plate.
  Arms: classical reduction and fixation

SUMMARY:
The aim of the current study was to evaluate the accuracy of computer-guided mandibular fracture reduction versus the classical work flow

DETAILED DESCRIPTION:
Research question:

Does the use of screw holes locating surgical guide & pre-bent plates osteosynthesis accurately reduce class III mandibular fractures regarding segments integrity and occlusion more than the classical reduction and fixation?

Statement of the problem:

Mandibular fractures are the most frequently occurring fractures within the maxillofacial injuries. The evaluation, diagnosis, and management of these fractures remain challenging despite improved imaging technology and fixation techniques. Depending on the type and location of the fractures, various open and closed surgical reduction techniques can be utilized. There are several critical and inherent limitations to the current ,standard approach of mandibular fracture reduction and fixation includes : (improper alignment of segments ,malocclusion ,nerve affections and related teeth roots injury).

There is a possibility to overcome these limitations with the help of computer-guided surgery . The introduction of CAD/CAM software has provided surgeons with an opportunity to perform virtual manipulations of CT datasets preoperatively and production of corrected mandibular model for plate pre-bending and fabrication of plate locating surgical guide which provide accurate segment reduction and fixation with accurate post-operative occlusion and minimal post-operative complication . The aim of the current study was to evaluate the accuracy of computer-guided mandibular fracture reduction versus the conventional work flow

Rationale for conducting the research:

Through computer guided mandibular fracture reduction investigators can provide proper segment alignment with subsequent accurate post-operative occlusion in addition reduce intra-operative time , post-operative pain and edema

ELIGIBILITY:
Inclusion Criteria:

* Patients with delayed and isolated mandibular class III fracture needs open reduction and internal fixation.
* Patients with medical history that did not hinder plate placement (uncontrolled diabetes) and adequate proper oral hygiene.
* Both genders males and females will be included.

Exclusion Criteria:

* • General contraindications to surgery.

  * Patients with fresh fractures (mobile segments).
  * Patients with unfavourable nor comminuted fractures.
  * Subjected to irradiation in the head and neck area less than 1 year before fixation.
  * Untreated periodontitis.
  * Poor oral hygiene and motivation.
  * Uncontrolled diabetes.
  * Pregnant or nursing.
  * Substance abuse.
  * Psychiatric problems or unrealistic expectations.
  * Severe bruxism or clenching.
  * Immunosuppressed or immunocompromised.
  * Treated or under treatment with intravenous amino-bisphosphonates.
  * Patients participating in other studies, if the present protocol could not be properly followed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
computer tomography | after 3 months
  the Computer Tomography Will calculate the segments deviation in mm. after 3 month .

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Omara, Study Director — Cairo University; mona el hadidy, Study Director — Cairo University

REFERENCES:
- [Derived] Gaber A, Hatem H, El M, Omara M. Precision of patient specific screw holes locating surgical guide and pre-bent plates osteosynthesis versus classical workflow in management of class III mandibular fracture. Maxillofac Plast Reconstr Surg. 2025 Dec 19;47(1):43. doi: 10.1186/s40902-025-00495-4. PMID 41417183
- See also: Reginald H.B. Goodday/Management of Fractures of the Mandibular Body and Symphysis. Oral Maxillofacial Surg Clin North Am. 2013 Nov;25 — https://pubmed.ncbi.nlm.nih.gov/24021623/
- See also: Evaluation of the Accuracy of Computer-Guided Mandibular Fracture Reduction. 2015 Jul;26(5):1587-91.doi: 10.1097/SCS.0000000000001773. — https://pubmed.ncbi.nlm.nih.gov/26163841/.
- See also: Parul Sinha , Gary Skolnick , Kamlesh B Patel , Gregory H Branham , John J Chi /A 3-Dimensional-Printed Short-Segment Template Prototype for Mandibular Fracture Repair. 2018 Sep 1;20(5):373-380 — https://pubmed.ncbi.nlm.nih.gov/29710318/
- See also: Comparison of 3D plate and locking plate in treatment of mandibular fracture-a clinical study. Oral Maxillofacial Surg 2017 Dec;21(4) — https://pubmed.ncbi.nlm.nih.gov/28785906/
- See also: Scott Lovald , Bret Baack, Curtis Gaball, Garth Olson, Anna 31 Hoard/Biomechanical optimization of bone plates used in rigid fixation of mandibular symphysis fractures. 2010 Aug — https://pubmed.ncbi.nlm.nih.gov/20537782/